CLINICAL TRIAL: NCT02179866
Title: SINGLE-CENTER, OPEN-LABEL, NON-RANDOMIZED STUDY INVESTIGATING THE EXCRETION BALANCE, PHARMACOKINETICS AND METABOLISM OF A SINGLE ORAL DOSE OF [14C]-LABELED RO5285119 IN HEALTHY MALE SUBJECTS
Brief Title: A Single-center Study to Investigate How Quickly and to What Extent a Radioactive Dose of RO5285119 is Absorbed, Metabolized and Eliminated From the Body of Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP29279; 2014-000277-40 (EudraCT Number)
Record Dates: First submitted 2014-06-11; First posted 2014-07-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (1):
- [14C]-labeled RO5285119 (Experimental): Single oral dose - drinking solution
  Interventions: Drug: RO5285119

INTERVENTIONS:
Drug: RO5285119 — Single oral dose of RO5285119 with approximately 2.1 MBq (56.6 uCi) [14C]-radiolabeled RO5285119 administered as a drinking solution under fasted conditions on Day -1

SUMMARY:
This study is designed to investigate the absorption, distribution, metabolism and elimination of a single oral dose of radiolabeled [14C]-labeled RO5285119 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants, 35 to 64 years of age, inclusive
* For men with a female partner of child-bearing potential: Agreement to use two methods of contraception, including one barrier method e.g. condom, during the treatment period and for at least 3 months after the last dose of study drug
* Participants who do not intend to donate sperm until at least 3 months after the last dose of the study drug

Exclusion Criteria:

* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis
* Any personal or familial history of seizures, epilepsy or other convulsive condition, previous significant head trauma, or other factors predisposing to seizures
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first dose administration
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to a subject
* History or presence of any clinically relevant ECG abnormalities, cardiovascular or cerebrovascular disease
* History of myopathy or muscle disorder
* History or evidence of any medical condition potentially altering the absorption, metabolism or elimination of drugs
* Any CYP3A inhibitor within 2 weeks or within 5 times the elimination half-life, whichever is longer, prior to dosing
* Any CYP3A inducer within 4 weeks or within 5 times the elimination half-life, whichever is longer, prior to dosing
* Infrequent bowel movements (less than once per 24 hours on average)
* Regular work with ionizing radiation or radioactive material

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactivity over time in urine and feces expressed as a percentage of the total radioactive dose administered | Up to Day 17
Pharmacokinetic profile of total drug-related material, RO5285119 and its metabolites, as appropriate in plasma, estimated Cmax | Up to Day 17

SECONDARY OUTCOMES:
Percent of dose recovered as total radioactivity, i.e. relative abundance of RO5285119 and its metabolite(s) in plasma, urine and feces | Up to Day 17
Incidence of adverse events | Up to 28 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands